CLINICAL TRIAL: NCT01748032
Title: The Effects of Short-term Cognitive Training on Cognition and Mood Symptoms in Late-life Depression: A Pilot Study
Brief Title: Short-term Cognitive Training in Late-life Depression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low Recruitment
Sponsor: Rotman Research Institute at Baycrest (Other)
Collaborators: Baycrest (Other)
Responsible Party: Principal Investigator, Linda Mah, MD, Clinician Scientist, Rotman Research Institute at Baycrest
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12-28
Record Dates: First submitted 2012-12-10; First posted 2012-12-12 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Depression
Keywords: depression; intervention studies
MeSH Terms: conditions — Depression | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Alternative Uses Training (Other): In this task, subjects are asked to produce atypical and alternative uses for common daily objects.
  Interventions: Behavioral: Cognitive training
- Word Association Training (Other): In this task, subjects are asked to generate the first word that comes to their mind, and thus, encourages more general and spontaneous divergent thinking.
  Interventions: Behavioral: Cognitive training

INTERVENTIONS:
Behavioral: Cognitive training — 20 minutes/day for 5 sequential working days
  Other Names: cognitive intervention

SUMMARY:
The purpose of this study is to examine the effects of the alternative uses training (AUT) and word association training (WAT) on cognitive functions and mood symptoms in late-life depression (LLD).

The hypotheses are:

1. post-training cognitive performance will be superior to pre-training cognitive performance
2. post-training depressive symptomatology will be less severe as compared with pre-training clinical severity and
3. AUT group will show better post-training cognitive performance and improved mood symptoms when compared with the WAT group.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age >=55
* Proficiency in English
* Current depressive episode and meet criteria for DSM-IV major depressive disorder
* Hamilton Depression Rating Scale score >=15
* Able to give informed consent
* Stable medication dosages during the training period

Exclusion Criteria:

* Other DSM-IV Axis I psychiatric disorders, except for anxiety disorders due to high comorbidity with mood disorders
* Mini-Mental State Examination score of <26
* Diagnosis of dementia
* Neurological and medical conditions known to affect cognition (e.g., stroke, head injury, previous chemotherapy for cancer)
* Unstable medical illnesses requiring active treatment
* Vision or hearing impairment affecting ability to participate in training

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-08; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Changes in cognitive functions including fluid intelligence, executive function, language, memory and motor speed | Within 3 days before the first cognitive training day and within 3 days after the last cognitive training day
  Computerized Executive Tasks:
  * Number-Letter Task
  * Letter-Memory Task
  * Stroop Task
  Non-Computerized Measures:
  * Cattell Culture Fair Intelligence Test
  * Mattis Dementia Rating Scale-2 (DRS-2)

SECONDARY OUTCOMES:
Changes in mood including depression, anxiety and apathy | Within 3 days before the first cognitive training day and within 3 days after the last cognitive training day
  * Montgomery Asberg Depression Rating Scale (MADRS)
  * Apathy Evaluation Scale (AES)
  * Hamilton Anxiety Rating Scale (Ham-A)
  * Beck Depression Inventory (BDI)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Mah, MD, M.H.Sc., Principal Investigator — Rotman Research Institute at Baycrest
Locations (1):
- Rotman Research Institute at Baycrest, Toronto, Ontario, Canada